CLINICAL TRIAL: NCT05464199
Title: Home-based EEG Neurofeedback to Reduce Chronic Neuropathic Pain, a Cohort Clinical Trial.
Brief Title: Home-based EEG Neurofeedback for Chronic Neuropathic Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: East Kent Hospitals University NHS Foundation Trust (Other Government)
Collaborators: Exsurgo Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022/NEURO/02
Record Dates: First submitted 2022-06-27; First posted 2022-07-19 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Neuralgia
Keywords: Neurofeedback
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Intervention Model Description: Single cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants receiving neurofeedback intervention (Experimental): Self administered neurofeedback training - Use of Headset and tablet with software App for playing a selected neurofeedback game. The EEG headset and tablet-based application is designed with the purpose of alleviating chronic pain by providing the user with feedback of, and allowing them to modulate, their own EEG signals associated with activity in brain networks related to pain perception and pain modulation.
  Interventions: Other: Neurofeedback training

INTERVENTIONS:
Other: Neurofeedback training — Self-administered neurofeedback treatment using headset and tablet-based application, designed with the purpose of alleviating chronic pain by providing the user with feedback of, and allowing them to modulate, their own brain EEG signals associated with activity in brain networks related to pain perception and pain modulation.
  Visual feedback will be provided onscreen representing the participant's real time EEG activity measured by the headset. Each session will be split into five blocks of five minutes each, with a one-minute rest period in between, in order to avoid fatigue and allow the participant to move around and adjust their position. After each rest block, participants will be asked if they are ready to proceed and when ready, the next block can be started. After the end of the session (5 blocks) the participant will then be asked to perform a post-session eyes-open EEG recording, similar to the eyes-open baseline taken at the start of the session.

SUMMARY:
In order to address the growing problem of chronic pain management in the UK, a proof of concept/feasibility open label cohort study has been devised to explore the effectiveness of a home-based self-administered non-pharmacological treatment utilising neurofeedback (NFB) training with a headset and tablet-based software application. This study will replicate the intervention from a previous clinical trial conducted in the UK during the Covid-19 lockdown in 2020/21 (NCT04418362) and extend it by examining EEG activity before, during, and after the intervention, alongside outcome measures, including changes in pain intensity and severity, sleep, mood and quality of life.

Ten participants will take part in pre-intervention assessments followed by four weeks of EEG baseline readings (5 times per week for 5 minutes), eight weeks of NFB treatment (5 times per week for 40 mins), and 12 weeks of post treatment EEG baselines readings (5 times per week for 5 minutes). Participants will be provided with training and detailed instructions on how to self-administer the NFB treatment using a bespoke headset and tablet-based software application in the comfort of their own homes.

Assessments will be conducted at Week 0 (pre-intervention), Week 4 (pre-NFB treatment), Week 12 (post NFB treatment) and at follow up points (Week 16, 20, and 24). It is anticipated this study will provide evidence of the safety, efficacy, reliability and validity of a low-cost non-pharmacological solution to the physical, psychological and social difficulties experienced by individuals with chronic neuropathic pain conducted within the NHS health system.

DETAILED DESCRIPTION:
This research trial aims to explore the feasibility, safety and effectiveness of an 8-week home-based EEG neurofeedback training programme for a sample of 10 individuals living with severe chronic neuropathic pain within the NHS treatment framework.

Neurofeedback training aims to modulate brain EEG activity arising from cortical and sub-cortical areas of the brain associated with pain perception and modulation, and preliminary findings suggest it could be a safe and effective tool in the treatment of chronic pain.

Several studies indicate that neurofeedback which aims to upregulate alpha frequency activity over sensorimotor areas of the brain can produce substantial improvements in pain. Recent systematic reviews have called for more robustly designed trials in terms of methodology and feasibility and for changes in EEG activity to be measured and correlated with outcome measure assessments.

A recent proof of concept study (Number of participants=16) was conducted in the UK during the Covid pandemic lockdown in 2020/21, to examine the safety and efficacy of a home-based EEG neurofeedback intervention for the management of chronic pain and associated symptoms. This study as referred to below, showed significant improvements in pain, central sensitisation, sleep, mood and quality of life measures for many of the heterogenous group, alongside correlations with changes in EEG activity.

Study title: Brain Train for Pain - A home-based neurofeedback intervention to treat the primary and secondary symptoms of chronic pain.

REC reference: 20/NW/0209 Protocol number: ED1001033 IRAS project ID: 277936

This trial will utilise an updated version of the equipment (Headset, tablet and software App) and replicate the neurofeedback intervention while expanding on the above study by showing changes in EEG activity during and after the intervention period in a homogenous cohort of participants living with chronic neuropathic pain. Furthermore, it will validate the efficacy of a home-based telehealth intervention for chronic neuropathic pain within the NHS.

The primary hypotheses of this study are that:

i) 8 weeks of usual care plus active EEG neurofeedback is feasible, safe, and clinically efficacious, resulting in a reduction in perceived pain, and improvement in central sensitisation, mood, sleep, and quality of life measures ii) Baseline EEG resting state activity will differ over three time points - pre, during, and post-intervention.

iii) Changes in EEG activity will be correlated with changes in primary and secondary outcome measures

The research team will conduct a simple single arm cohort study measuring outcomes before and after an 8-week period of neurofeedback intervention and then throughout a follow up period of 12 weeks. The total time period for each participant will be 23 weeks.

All potential applicants will be screening against eligibility criteria. Individuals who meet the eligibility criteria will be invited to take part in this trial.

Potential participants will be recruited from a variety of sources including East Kent Hospitals University NHS Foundation Trust (EKHUFT) Out-patient clinics (primarily from the Out-patient clinic of the Chief Investigator), patient association networks (for example: Kent Multiple Sclerosis Therapy Centre and Headway Kent), NHS primary care in East Kent and social media may also be used.

Participant time-line -

Week 1 - EEG baseline measurements (5 times during the week for 5 mins) and initial outcome measurements Week 2 - Transition week - Research team video based appointment for checking all aspects and further training required and outcome measure assessment.

Weeks 3 to 10 - active self administered neurofeedback treatment by participant at home - 5 times per week for 40 minute sessions.

Weeks 11 to 23 - EEG baseline measurements (5 times per week for 5 mins). 4 video based follow up appointments with a member of the research team for outcome measurements and checking and confirmation of any potentially reported issues.

After completion of the trial, all participants will be provided with a debrief document to enable participants to have an opportunity to discuss anything they would like with the Chief Investigator and also to enable them to have the opportunity of obtaining a brief 1-page summary report of the results of the research after all data and results have been analysed.

Statistical Analysis.

Study results will first undergo descriptive level statistical analyses. Continuous variables will be reported using mean (standard deviation) or median (interquartile range), depending on the data distribution, and dichotomous and categorical variables will be reported using frequencies (proportion). All data will be analysed following intention-to-treat principles. Secondary per protocol analyses may also be completed. The difference in primary and secondary outcomes will be analysed with linear or general linear mixed effects models, controlling for baseline scores. The research team will report the number of participants with missing scores for each outcome and any imputations will be carried out consistent with the approaches laid out in Gelman and Hill (Ref: Gelman A. and J. Hill, Missing-data Imputation in Data Analysis Using Regression and Multilevel/Hierarchical models. 2006, London, UK. p. 529-544.)

The research team will report imputation methods, and will perform a sensitivity analysis, examining effects on the outcomes reported, using the approach recommended by White et al (Ref: White, I.R., et al., Strategy for intention to treat analysis in randomised trials with missing outcome data. BMJ, 2011. 342: p. d40.)

For the secondary outcome measures, linear mixed effects models will also be used to assess the relationship between % improvement in Brief Pain Inventory and Visual Analogue Scale for pain average changes 1) in resting EEG alpha frequency band power, relative alpha, hi-beta and theta, pre to post intervention and at all follow up points. Potentially important covariates (e.g. baseline pain intensity, psychological distress, sleep quality) will also be assessed for interaction, collinearity and confounding. With respect to participant safety, discontinuation rates, adverse events and treatment emergent adverse events will all be reported and documented.

ELIGIBILITY:
Inclusion Criteria:

* Males and females over 18 years of age with ongoing chronic neuropathic pain for 3 months or more
* must have had an average pain rating in the last week of equal to or greater than 4/10 on Visual Analogue Scale for Pain
* must have a head circumference between 520-620 mm to ensure correct fitment of headset
* must have access to a reliable internet connection and Wi-Fi at home
* must have and display competence with equipment and headset usage after training

Exclusion Criteria:

* Previous neurofeedback training
* serious recent (within 12 months) head injury and/or traumatic brain injury and/or concussion
* diagnosed with a major neurological disorder (e.g. trigeminal neuralgia)
* a history of seizures
* diagnosed with a major psychiatric disorder
* has an implanted electronic neuromodulation device for example - a heart pacemaker, or loop recorder
* is unable to provide informed consent
* must not have any change in medication or treatment planned in the 1 week prior to and during the trial intervention period, or in the 12 weeks post trial intervention, while EEG baselines are being recorded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-08-16 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Pain Scale | 23 weeks
  Unidimensional measure of pain intensity - Numeric scale from 0 (no pain) to 10 (worst pain ever). Number is chosen by participant to rate their pain.
Brief Pain Inventory | 23 weeks
  A self-reported scale that measures the frequency, and severity of pain and the interference of pain on various domains of daily activity. The severity items ratings range from 0 (no pain) to 10 (pain as bad as you can imagine).

SECONDARY OUTCOMES:
Depression Anxiety and Stress Outcome Scale 21 | 23 weeks
  Self rated scale on depression anxiety and stress
Pain Catastrophizing Scale | 23 weeks
  Self rated scale on perception of pain
Central Sensitization Inventory | 23 weeks
  Self rated scale used to determine central sensitisation to pain
Pittsburg Sleep Quality Index | 23 weeks
  Self rated scale on sleep
Health related perceived quality of life EuroQol scale | 23 weeks
  Self rated scale on perceived health related quality of llife
Brain Electroencephalogram EEG recordings | 23 weeks
  Objective changes in individual brain EEG recordings - Alpha, Beta and Theta Wavelengths

CONTACTS AND LOCATIONS:
Overall Officials: Dr Mohamed Sakel, MBBS, Principal Investigator — East Kent Hospitals University NHS Foundation Trust
Locations (1):
- East Kent Hospitals University NHS Trust, Canterbury, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sakel M, Ozolins CA, Saunders K, Biswas R. A home-based EEG neurofeedback treatment for chronic neuropathic pain-a pilot study. Front Pain Res (Lausanne). 2025 Mar 11;6:1479914. doi: 10.3389/fpain.2025.1479914. eCollection 2025. PMID 40134759